CLINICAL TRIAL: NCT00317668
Title: Role of Antibodies Against Glutamate Receptors and Double Stranded DNA in Epilepsy Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: autoimmunepi-HMO-CTIL
Record Dates: First submitted 2006-04-23; First posted 2006-04-25 (Estimated); Last update posted 2007-05-01 (Estimated); Status verified 2006-04

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The investigators will check the serum of epilepsy patients for antibodies against glutamate receptors and double stranded DNA. They will characterise the patients (by the kind of epilepsy, autoimmune disease comorbidity, and cognitive profile).

ELIGIBILITY:
Inclusion Criteria:

* 120 epilepsy patients from the epilepsy clinic and Emergency Room (ER)
* Controls: 100 patients with other neurological diseases and no epilepsy; and 30 healthy volunteers.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2006-11

CONTACTS AND LOCATIONS:
Overall Officials: Dana Ekstein, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Ein-Kerem Medical Center, Jerusalem, Israel